CLINICAL TRIAL: NCT06779032
Title: Clinical Profile of Skin Aging Based on Dermoscopy Photoaging Scale and Glogau Scale - Study of Leucocyte Telomere Length, Biomarker P16, and Body Mass Index
Acronym: LTLP16
Status: Not yet recruiting | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, Sp.DVE, Subsp. D.K.E, Indonesia University
Other Study IDs: LTLP16
Record Dates: First submitted 2024-12-22; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Aging Skin; Body Mass Index; Cellular Senescence; Triglycerides; Waist Circumference
Keywords: skin aging; body mass index; triglycerides; waist circumference; cellular senescene; p16
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- leucocyte telomere length (LTL): patients will be assessed LTL to see if there is correlation with body mass index, triglycerides, and skin aging
  Interventions: Diagnostic Test: blood draw
- p16: patients will be assessed p16 to see if there is correlation with body mass index, triglycerides, and skin aging
  Interventions: Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: blood draw — PCR method to see leucocyte telomere length
Diagnostic Test: blood draw — PCR method to see p16

SUMMARY:
To determine the relationship between clinical appearance, dermoscopic examination results of photoaging profiles based on clinical examination, DPAS score and leucocyte telomere length, to analyze the relationship between BMI, waist circumference, triglycerides, and cellular senescence biomarker p16 levels with a population experiencing skin aging and having Fitzpatrick III-V skin types.

The questions which is aim to be answered are:

1. What is the photoaging profile based on clinical examination results in skin aging cases?
2. What is the photoaging profile based on DPAS scores in skin aging cases?
3. What is the leucocyte telomere length profile in skin aging cases?
4. What is the relationship between leucocyte telomere length and clinical examination in skin aging cases?
5. What is the relationship between leucocyte telomere length and DPAS degree in skin aging cases?
6. What is the profile of cellular senescence p16 biomarker levels in a population that has experienced clinical skin aging with Fitzpatrick III-V skin types?
7. What is the skin aging profile based on the Glogau and DPAS scales in a population with Fitzpatrick III-V skin types?
8. Is there a relationship between the results of the cellular senescence p16 biomarker examination and clinical skin aging assessed based on the Glogau and DPAS scales in a population with Fitzpatrick III-V skin types?
9. Is there a relationship between the results of BMI, waist circumference, and triglyceride examinations with clinical skin aging assessed using the Glogau and DPAS scales with Fitzpatrick III-V skin types?

DETAILED DESCRIPTION:
Skin aging is a process of decreasing the structure and physiological function of the skin that significantly increases in the 4th and 5th decades of age. The skin is the largest organ which is one-sixth of the total body weight in humans. One of the functions of the skin is as a protective organ that borders the external environment of the body, therefore, indicators of aging can be clearly seen on the skin. Some clinical manifestations of photoaging are wrinkles, rough, dry skin, telangiectasis, precancerous lesions, and changes in skin pigmentation. Photoaging assessment was first proposed in 1996 by Dr. Richard Glogau. The Glogau scale assesses photoaging based on clinical assessments which are grouped into 4 categories, namely types I, II, III, and IV. There is no literature on the validity and reliability of the Glogau scale, especially in individuals with Fitzpatrick skin types III and IV. Asian populations, especially those with Fitzpatrick skin types III, IV, and V, tend to experience pigmentation problems such as post-inflammatory hyperpigmentation and melasma. A study by Du et al found that Indonesian women, in particular, consider pigmentation and skin color imbalance as a major problem. Skin aging problems can affect patients' self-confidence and quality of life, although they are not life-threatening. The number of skin aging cases increased from 4.8% in 2021 to 11.5% in 2023, according to outpatient visit data at the Cosmetic Dermatology Polyclinic, KSM Dermatology and Venereology (DV) FKUI-RSCM. Along with the development of medical technology, in 2013 a photoaging evaluation instrument using dermoscopy was created, namely the dermoscopy photoaging scale (DPAS). The study was conducted in Istanbul with research subjects who mostly had Fitzpatrick skin types II and III. Dermoscopy findings assessed are manifestations of clinical photoaging such as skin discoloration, skin atrophy, telangiectasis, actinic keratosis, senile comedones, and wrinkles. The score is calculated based on specific dermoscopic findings in 4 facial regions, namely the forehead, chin, and both cheeks, which are then added up to a maximum score of 44. Dermoscopic evaluation as a simple and non-invasive diagnostic tool is more objective than clinical assessment. Assessment using DPAS is easy to use, can be applied in various situations and the score can be calculated quickly. Dermoscopic examination results will be compared with leucocyte telomere length (LTL) examination. Telomere shortening can cause cell aging, and from various studies, this has been studied as a marker of aging and a risk factor for age-related diseases. Telomere shortening accelerates skin aging. Clinically, skin aging is associated with reduced skin barrier function, poor wound healing, increased inflammation, disturbed water and temperature homeostasis, and increased susceptibility to skin disorders, including skin cancer. The main characteristics of aging, which are found in all parts of the body, are interconnected with each other, characterized by progressive loss of physiological integrity, genome instability, decreased telomere length, epigenetic changes, loss of proteostasis, decreased nutrient regulation, mitochondrial dysfunction, cellular senescence, stem cell exhaustion, and impaired intercellular communication.

Cellular senescence is considered one of the main characteristics of aging, which is defined as a growth arrest mediated by cell cycle regulators p53, p21, and p16. P16, has an important role in controlling the retinoblastoma tumor suppressor protein. Senescent cells that are positive for p16 accumulate in aging tissues including the skin.

The lack of clarity in the results of the correlation between p16 and skin aging assessed clinically using the Glogau scale and dermoscopy with the DPAS scale, has encouraged researchers to conduct a study to see the results of the levels of these cellular aging biomarkers in the Indonesian population. The results of the study are also expected to be able to correlate the p16 biomarker with clinical skin aging experienced at various ages in men and women. Several factors such as body mass index (BMI), waist circumference, triglycerides, can affect skin aging. A person with overweight or obese BMI has a changed skin structure compared to a person with normal BMI. People with obesity have a less well-organized skin collagen structure caused by degradation of collagen fibers and these dermal changes are irreversible. In obesity, skin-resident and systemic adipose tissue secrete several factors and increase inflammation and have a detrimental effect on facial aging.

Waist circumference is part of the adiposity indicator parameters other than BMI. Facial aging is related

ELIGIBILITY:
Inclusion Criteria:

* female aged 31-61 years
* healthy
* willing to participate in the study

Exclusion Criteria:

* history of diseases (heart, kidney, liver)
* pregnant or breastfeeding patientes

Ages: 31 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: people with age from 31- 61 years
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
profile of leucocyte telomere length | 1 year
  profile of leucocyte telomere length in skin aging
profile of skin examination with dermoscopic photoaging scale (DPAS) | 1 year
  skin aging is assessed from dermoscopic photoaging scale on dermoscopic images, looking at pigmentary changes, vascular changes, telangiectasis, wrinkles, actinic keratoses, and blackheads. There are four facial regions assessed in the DPAS score calculation, namely the forehead, right cheek, left cheek, and chin. The sum of the scores of the four regions is assessed based on 11 parameters, with a maximum final score of 44.
  The greater the score, the higher marks of skin aging
Profile of body mass index | 1 year
  checking BMI to see if there is correlation so skin aging
profile of p16 | 1 year
  checking p16 as a cellular senescence to skin aging
profile of waist circumference | 1 year
  Waist circumferemce will be checked, to see if there is correlation with skin aging
profile triglycerides | 1 year
  triglycerides will be checked, to see if there is correlation with skin aging

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided